CLINICAL TRIAL: NCT07254429
Title: Copenhagen Menopause Study (COMPASS): A Randomized Clinical Trial
Brief Title: COMPASS - COpenhagen MenoPAuSe Study
Acronym: COMPASS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Professor, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-522558-37-00; 2025-522558-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-30; First posted 2025-11-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Menopausal Osteoporosis; Bone Markers
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Triptorelin Pamoate; Sodium Chloride; Estradiol; Testosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GnRH analog (Active Comparator): Pamorelin 11.25 mg intramuscular injection once + Daily placebo gel
  Interventions: Drug: Triptorelin 11.25 mg; Drug: Placebo gel
- Placebo (Placebo Comparator): Saline intramuscular injection once + Daily placebo gel
  Interventions: Drug: Sodium Chloride 0.9%; Drug: Placebo gel
- Transdermal Estrogen (Active Comparator): Saline intramuscular injection once + Estreva gel 1.5 mg daily
  Interventions: Drug: Sodium Chloride 0.9%; Drug: Estradiol (E2)
- Transdermal testosterone (Active Comparator): Saline intramuscular injection once + Tostran gel 10 mg every other day + placebo gel every other day
  Interventions: Drug: Sodium Chloride 0.9%; Drug: Testosterone; Drug: Placebo gel

INTERVENTIONS:
Drug: Triptorelin 11.25 mg — Pamorelin 11.25 mg intramuscular injection once
  Other Names: Pamorelin
  Arms: GnRH analog
Drug: Sodium Chloride 0.9% — Saline intramuscular injection once
  Other Names: Saline
  Arms: Placebo; Transdermal Estrogen; Transdermal testosterone
Drug: Estradiol (E2) — Estreva gel 1.5 mg daily
  Other Names: Estreva
  Arms: Transdermal Estrogen
Drug: Testosterone — Tostran gel 10 mg every other day
  Other Names: Tostran
  Arms: Transdermal testosterone
Drug: Placebo gel — Placebo gel every day or every other day
  Arms: GnRH analog; Placebo; Transdermal testosterone

SUMMARY:
During menopause, estrogen levels drop while the level of another hormone - LH (luteinizing hormone) substantially increases. This hormonal shift is linked to bone Loss and other complications. Estrogen therapy can help, but some women avoid it due to the increased risk of blood clots and cancer. This project will investigate whether blocking LH could offer a safe alternative to alleviate symptoms and complications of menopause since it is known from previous research that high LH levels contribute to both bone deterioration and metabolic issues. The goal is to explore new treatment options that can improve health and quality of life for women both during and after menopause. This randomized clinical trial is a single center, sponsor-investigator-initiated single-blinded 8 weeks clinical trial with four parallel groups comparing the effect of an gonadotropin releasing hormone(GnRH)-analog with placebo, and with two additional arms given estrogen or testosterone on change on bone health in postmenopausal women with moderate-to-severe symptoms.

DETAILED DESCRIPTION:
The hormonal changes occurring in perimenopause and menopause exert multiple effects on several organs and the accompanied symptoms can be very distressing and impair quality of life. Vasomotor symptoms (VMS) defined as hot flashes and sweating are the most frequent and bothersome symptoms of menopause and are experienced by up to 80% of women. Additionally, in the Western world, 66% of postmenopausal women are obese and 54% have osteoporosis. Along with obesity comes a wide variety of health issues such as type 2 diabetes, metabolic syndrome, and atherosclerosis, which can lead to cardiovascular disease. Osteoporosis is a huge economic cost for society, it impairs quality of life and vertebral and hip fractures are associated with increased mortality. Postmenopausal symptoms and complications take a large toll on both the physical and mental well-being of women and are a huge cost to society. Menopausal Hormonal Therapy (MHT) with estrogen and gestagen is used by many women as it alleviates symptoms and reduces the risk of osteoporosis and cardiovascular disease. However, due to the increased risk of breast cancer and venous thromboembolism, some women refuse MHT and there is an ongoing search for new treatments. The newly approved Veoza® (Fezolinetant) is also approved and on the marked, but only targets VMS and not menopausal complications, but can be a treatment option, if the woman can or will not have MHT.

Menopause is characterized by low circulating estrogen, but also by very high levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH), and these hormonal changes are linked with increased bone resorption and weight gain. Despite the high LH in menopause, LH pulses occur simultaneously with hot flashes also in postmenopausal women, and LH may be involved in the events. In a clinical study 10 postmenopausal women with severe VMS were given a GnRH antagonist cetrorelix 250 μg two times a day in 6 weeks. They found a significant decrease in VMS symptoms. Postmenopausal women experience a decline in core temperature, which we suggest is due to LH actions on brown and white fat cells leading to less heat generation, beta-oxidation, and more storing of fat. Furthermore, LH appears to be a rapid and potent inducer of renal calcium excretion, which induces a secondary and persistent increase in parathyroid hormone (PTH) that mobilizes calcium from the skeleton. The LH-induced calcium excretion occurs several hours before the subsequent changes in sex steroids, particularly estrogen, which indicates a direct effect of LH that can lead to increased bone resorption and eventually osteoporosis. This may be of great importance during the perimenopause/early phase of menopause, where the decrease in bone mineral density and increase in visceral adiposity is high concurrent with serum LH increasing dramatically, while serum estrogen is still not greatly reduced. The investigators propose to investigate if lowering LH using a gonadotropin releasing hormone (GnRH) analog against placebo can improve bone markers and secondarily reduce the frequency and severity of VMS in postmenopausal women with a direct comparison to estrogen - the gold standard treatment of women in menopause, and testosterone in the same RCT.

The main aim of the study is to show that by targeting LH the investigators can change bone markers and maybe even combat hot flashes and night sweats (VMS) in postmenopausal women. For important biological knowledge purpose, the investigators also investigate the 2 additional treatment arms with estradiol and testosterone to compare the effect against the current gold standard treatment option (estradiol) and to testosterone, which is a common supplement to postmenopausal women off-label. A study by Glaser et al. effectively documents that testosterone can improve most common post-menopausal symptoms.

Sample size calculation and statistics Previous studies have shown that CTX in postmenopausal women is usually between 0.44 ng/mL with a standard diviation on SD 0.2. The sample size is calculated based on a direct comparison between GnRH analog (pamorelin) and placebo on the primary outcome 'change in bone markers' (delta CTX between pamorelin and placebo), using a power of 80% and alpha of 0.05 leads to 44 participants in each group, and the investigators would be able to detect a change in CTX on 30 %. The calculations is based on only two arms, however for comparison reasons the investigators will include two extra arms with estradiol/testosterone and patients will be allocated 1:1:1:1 leading to a total sample size of 176 participants. Our design and analysis principles rely on the intent-to-treat (ITT) approach; the investigators strive to evaluate and include all randomized participants in the primary analysis, regardless of adherence to treatment assignment or protocol requirements.

The investigators estimate to screen 250 to include 192 to be randomized and 176 to complete the study leaving 16 patients for dropout (9%). The design enables us to investigate multiple secondary outcomes where the primary comparison will be between GnRH analog treatment and placebo. The study is not powered to show significant differences between placebo and GnRH treatment for most secondary endpoints and should be considered as a pilot placebo-controlled intervention study for these outcomes. T-tests will be used for the primary endpoint, while Nonresponder imputation will be used for missing response data. Change in mean frequency and severity of VMS per 24 hours will be analyzed for each week using a mixed effect model for repeated measures, with change from baseline as the dependent variable and treatment group, visit, and smoking status as factors and baseline measurement as a covariate, as well as interaction of treatment by week and an interaction of baseline measurement by week.

Predefined subgroups: Efficacy in patients with detectable versus undetectable serum hCG, high versus low LH at baseline, low versus high BMI, low versus high BMD, low versus high fat %.

Ethics and side effects All patients will be informed of potential adverse effects, and that they can leave the trial at any point without any consequences. GnRH-analogs have been proven safe in numerous randomized clinical trials (RCT) and have for many years been involved in the treatment of several groups including children with precocious puberty, transgender hormone treatment, and as part of in vitro fertilization. MHT have been tested in previously large RCT, where an increased risk of breast cancer and thromboembolic events have been detected. It is estimated that the risk of breast cancer increases with 0.5 % after 5 years of hormonal treatment. It is therefore regarded safe for participant in this trial to be treated with estrogen in 8 weeks however women with increased risk of cancer or thromboembolic events will be excluded. All side effects will be closely monitored and reported. The study will be approved by the regional ethical committee, conducted in compliance with The Declaration of Helsinki, registered on clinicaltrial.gov, and monitored by the GCP unit of Copenhagen University Hospitals in compliance with International Conference on Harmonisation.

ELIGIBILITY:
Inclusion Criteria:

* Women >40 years and ≤65 at screening visit
* A body mass index between 18-35
* Confirmed menopause

  * Method 1
  * Spontaneous amenorrhea for ≥12 consecutive months
  * Negative urine hCG test
  * Method 2
  * Spontaneous amenorrhea for ≥6 months
  * FSH >30 mIU/L
  * Negative urine hCG test
* Moderate to severe vasomotor symptoms (VMS)

  * Within the 7 days prior to randomization, participants must report ≥ 14 moderate to severe VMS per week

Exclusion Criteria:

* Current or previous hormone replacement therapy (HRT)

  * Vaginal estradiol/vaginal inserts (e.g. Vagifem®) can be used, but will have to be pause 2 weeks prior to randomization and throughout the study period
  * Menopausal Hormone Therapy (MHT) can be used by participants, but must be paused 6 weeks prior to inclusion.
* Current or previous cancer diagnosis

  * Except for basal cell carcinoma
* Known BRCA gene mutation
* Current hyperthyroid disease
* Osteoporosis
* Major psychiatric diagnosis including ongoing medication e.g. selective serotonin re-uptake inhibitors (SSRIs)
* Known prolonged QT or other known clinically significant abnormal ECG, including taking medication that can prolong QT interval (e.g. sotalol, dronedarone, amiodarone, methadone, and several antipsychotic drugs)
* Previous myocardial infarction or heart failure
* Previous thromboembolic event
* The use of opioids, anticoagulating treatment or unwilling to pause fish oil/Omega-3 supplements 3 days prior visit 1 and 3
* Current alcohol or drug abuse
* Hypertension treated with more than two drugs
* Severe history of allergy, hypersensitivity, or intolerance to drugs
* Moderate to severe liver and kidney disease (eGFR <60 mL/min)
* Diagnosed with type 1 or 2 diabetes
* Chronic diseases requiring immunomodulatory treatments such as rheumatoid arthritis, inflammatory bowel disease, and vasculitis etc.
* Known uterine fibroids, Endometriosis, Systemic lupus erythematosus (SLE), otosclerosis, severe migraine or sleep apnea
* Known Epilepsy or previous seizures or convulsive disorder

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in bone remodeling from baseline to week 8. | From baseline to week 8
  Change in bone remodeling defined by change in bone marker (ΔCTX) from baseline to week 8.
  The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between:
  1. GnRH analog and placebo-group.
     After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order:
  2. Combined analysis of all 4 arms of the RCT
  3. GnRH analog and estradiol
  4. GnRH analog and testosterone
  5. Estradiol and placebo
  6. Testosterone and placebo
  7. Estradiol and testosterone
Change in bone remodeling from baseline to week 8. | From baseline to week 8
  Change in bone remodeling defined by change in bone marker (ΔP1NP) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in bone remodeling from baseline to week 8 | From baseline to week 8
  Change in bone remodeling defined by change in bone marker-ratios (ΔCTX/ΔP1NP, and ΔBBI) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone

SECONDARY OUTCOMES:
Change in serum levels of Hypothalamic-Pituitary-Adrenal (HPA) axis from baseline to week 8 | Baseline to week 8
  Change in serum levels of Hypothalamic-Pituitary-Adrenal (HPA) axis from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum levels of Hypothalamic-Pituitary-Gonadal (HPG) axis from baseline to week 8 | Baseline to week 8
  Change in serum levels of Hypothalamic-Pituitary-Gonadal (HPG) axis from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum levels of Hypothalamic-Pituitary-Thyroid (HPT) axis from baseline to week 8 | Baseline to week 8
  Change in serum levels of Hypothalamic-Pituitary-Thyroid (HPT) axis from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in quality of life evaluated with MENQOL-1 from baseline to week 8 | Baseline to week 8
  Change in quality of life evaluated with The Menopause-specific Quality of Life (MENQOL) Questionnaire from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. MENQOL is ranging from 0 (asymptomatic woman) to 232 (extremely bothered).
Change in sexual function evaluated with female sexual function index from baseline to week 8 | Baseline to week 8
  Change in sexual function evaluated with female sexual function index (FSFI) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. The FSFI use a 5-point Likert scale with higher scores indicating greater levels of sexual functioning on the respective item. The possible range is 2-36.
Change in sexual function evaluated with female sexual distress scale-revised from baseline to week 8 | Baseline to week 8
  Change in sexual function evaluated with female sexual distress scale-revised (FSDS-R) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. FSDS-R has a total score ranging from 0 to 52, with higher scores indicating more sexually related distress.
Change in depressive symptoms evaluated by MDI from baseline to week 8 | Baseline to week 8
  Change in depressive symptoms evaluated by Major Depression Inventory (MDI) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Total score between 0 (no depression) to 50 (maximum depressed).
Change in depressive symptoms evaluated by CES-D from baseline to week 8 | Baseline to week 8
  Description: Change in depressive symptoms evaluated by Center for Epidemiologic Studies Depression Scale (CES-D) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Change in anxiety symptoms evaluated by GAD-7 from baseline to week 8 | Baseline to week 8
  Change in anxiety symptoms evaluated by General Anxiety Disorder-7 (GAD-7) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Scores ranges from 0 (No anxiety) to 21 (severe anxiety).
Change in The Mean Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b) from baseline to week 8 | Baseline to week 8
  Change in The Mean Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Scores ranges from 8-40. Higher scores indicate more severe sleep disturbance.
Change in thyroid hormones from baseline to week 4 and 8 | Baseline to week 4 and 8.
  Change in thyroid hormones from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine calcium from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in urine calcium from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine creatinine from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8.
  Change in urine creatinine from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine phosphate from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in urine phosphate from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine magnesium from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in urine magnesium from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine sodium from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in urine sodium from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in urine cortisol and other hormones from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8.
  Change in urine cortisol and other hormones from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum ionized calcium from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum ionized calcium from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum calcium from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum calcium from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum albumin from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum albumin from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum PTH from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum PTH from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum phosphate from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum phosphate from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum vitamin D metabolites from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum vitamin D metabolites from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum hCG from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum hCG from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in thyroid hormone conversion (DIO2 activity) in fat cells determined by their conversion of T4 to T3 from baseline to week 8 | Baseline to week 8
  Change in thyroid hormone conversion (DIO2 activity) in fat cells determined by their conversion of T4 to T3 from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in adrenal hormones from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in adrenal hormones from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in the mean frequency of moderate to severe VMS from Baseline to week 8 | Baseline to week 8
  Change in the mean frequency of moderate to severe VMS from Baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Definition of moderate VMS: Moderate VMS is defined as a sensation of heat with sweating/dampness, but the woman is able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Definition of severe VMS: Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity. If at night
Change in the mean frequency of moderate to severe VMS from Baseline to week 4 | Baseline to week 4
  Change in the mean frequency of moderate to severe VMS from Baseline to week 4. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Definition of moderate VMS: Moderate VMS is defined as a sensation of heat with sweating/dampness, but the woman is able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Definition of severe VMS: Severe VMS is defined as sensation of intense heat with sweating, caused disruption of activity. If at night
Change in the mean severity-score from Baseline to week 8 | Baseline to week 8
  Change in the mean severity-score from Baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Definition of mean severity-score of VMS: Severity score of moderate to severe VMS per day was calculated as follows: ((number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3))/Total number of daily hot flashes.
Change in the mean severity-score from Baseline to week 4 | Baseline to week 4
  Change in the mean severity-score from Baseline to week 4. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Definition of mean severity-score of VMS: Severity score of moderate to severe VMS per day was calculated as follows: ((number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3))/Total number of daily hot flashes.
Change in VMS measured by the Greene Climacteric Scale (GCS) from baseline to week 8 | Baseline to week 8
  Change in VMS measured using the questionnaire: The Greene Climacteric Scale (GCS) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Ranging from 0 (when every symptom is rated as "not at all") to a maximum of 63 (when every symptom is rated as "very often")
Change in serum LH from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in serum LH from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum FSH from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in serum FSH from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum estradiol from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum estradiol from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum SHGB from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum SHGB from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in physical strength tests from baseline to weeks 4 and 8. | Baseline to weeks 4 and 8.
  Change in physical strength test measured by 30 second Sit-To-Stand-Test (STST) from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. Unit: number of stands/30 seconds.
Change in physical strength tests from baseline to weeks 4 and 8. | Baseline to weeks 4 and 8.
  Change in physical strength test measured by Hand-grip strength (HGS) from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone. HGS will be evaluated using a digital hand-grip dynamometer measuring the absolute (kilograms-force) and relative (kilograms/weight in kilograms) grip strength

OTHER OUTCOMES:
Change in fasting insulin from baseline to week 8 | Baseline to week 8
  Change in fasting insulin from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in HbA1C from baseline to week 8 | Baseline to week 8
  Change in HbA1C (mmol/mol) from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in HOMA-IR from baseline to week 8 | Baseline to week 8
  Change in HOMA-IR from baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone.
Change in total cholesterol, cholesterol (total, HDL, LDL), and triglycerides from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in total cholesterol, cholesterol (total, HDL, LDL), and triglycerides from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum RANKL from baseline to weeks 4 and 8 | Baseline to weeks 4 and 8
  Change in serum RANKL from baseline to weeks 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum creatinine from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum creatinine from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum sodium from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum sodium from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum potassium from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum potassium from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in serum urea from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in serum urea from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in hepatic enzymes (ALAT, ASAT, GGT, alkaline phosphatase) from baseline to week 4 and 8 | Baseline to week 4 and 8
  Change in hepatic enzymes (ALAT, ASAT, GGT, alkaline phosphatase) from baseline to week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in QTc using electrocardiogram (ECG) at baseline to week 8 | Baseline to week 8
  Change in QTc using electrocardiogram (ECG) at baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in weight at baseline to week 8 | Baseline to week 8
  Change in weight at baseline to week 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in RNA expression (RNAseq) in abdominal fat (abdominal fat biopsies) from baseline to week 8 and following in vitro stimulation with hormones and treatments such as LH/hCG | Baseline to week 8
  Change in RNA expression (RNAseq) in abdominal fat (abdominal fat biopsies) from baseline to week 8 and following in vitro stimulation with hormones and treatments such as LH/hCG. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in Cerebral Spinal Fluid (CSF) hormone, mineral or neuropeptide levels between all 4 treatment arms at week 8 | between all 4 treatment arms at week 8
  Change in Cerebral Spinal Fluid (CSF) hormone, mineral or neuropeptide levels between all 4 treatment arms at week 8.
Change in frequency and type of reported adverse events between baseline and week 4 and 8 | Baseline and week 4 and 8
  Change in frequency and type of reported adverse events between baseline and week 4 and 8. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone
Change in ECG pattern from screening to week 4. | Screening to week 4.
  Change in ECG pattern from screening to week 4. The following primary, secondary and exploratory endpoints will all be investigated as comparisons first and foremost between: 1) GnRH analog and placebo-group. After the first analysis between GnRH-analog group and placebo, the outcomes will be investigated between the groups in the following order: 2) Combined analysis of all 4 arms of the RCT 3) GnRH analog and estradiol 4) GnRH analog and testosterone 5) Estradiol and placebo 6) Testosterone and placebo 7) Estradiol and testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Martin Blomberg Jensen, D.M.Sc., Principal Investigator — Herlev Hospital
Locations (1):
- Division of Translational Endocrinology, Department of Endocrinology and Internal Medicine, Copenhagen University Hospital Herlev., Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen HN, Moses AC, Garber J, Iloputaife ID, Ross DS, Lee SL, Greenspan SL. Serum CTX: a new marker of bone resorption that shows treatment effect more often than other markers because of low coefficient of variability and large changes with bisphosphonate therapy. Calcif Tissue Int. 2000 Feb;66(2):100-3. doi: 10.1007/pl00005830. PMID 10652955
- [Background] Langdahl B, Chung YS, Plebanski R, Czerwinski E, Dokoupilova E, Supronik J, Rosa J, Mydlak A, Rowinska-Osuch A, Baek KH, Urboniene A, Mordaka R, Ahn S, Rho YH, Ban J, Eastell R. Proposed Denosumab Biosimilar SB16 vs Reference Denosumab in Postmenopausal Osteoporosis: Phase 3 Results Up to Month 12. J Clin Endocrinol Metab. 2025 May 19;110(6):e1951-e1958. doi: 10.1210/clinem/dgae611. PMID 39243386
- [Background] Kline GA, Holmes DT. Bone turnover markers for assessment of anti-resorptive effect in clinical practice: A good idea meets the problem of measurement uncertainty. Clin Biochem. 2023 Jun;116:100-104. doi: 10.1016/j.clinbiochem.2023.04.007. Epub 2023 Apr 19. PMID 37084998
- [Background] Brown JP, Don-Wauchope A, Douville P, Albert C, Vasikaran SD. Current use of bone turnover markers in the management of osteoporosis. Clin Biochem. 2022 Nov-Dec;109-110:1-10. doi: 10.1016/j.clinbiochem.2022.09.002. Epub 2022 Sep 9. PMID 36096182
- [Background] Migliorini F, Maffulli N, Spiezia F, Peretti GM, Tingart M, Giorgino R. Potential of biomarkers during pharmacological therapy setting for postmenopausal osteoporosis: a systematic review. J Orthop Surg Res. 2021 May 31;16(1):351. doi: 10.1186/s13018-021-02497-0. PMID 34059108
- [Background] Everts-Graber J, Reichenbach S, Ziswiler HR, Studer U, Lehmann T. A Single Infusion of Zoledronate in Postmenopausal Women Following Denosumab Discontinuation Results in Partial Conservation of Bone Mass Gains. J Bone Miner Res. 2020 Jul;35(7):1207-1215. doi: 10.1002/jbmr.3962. Epub 2020 Feb 11. PMID 31991007
- [Background] Tsourdi E, Langdahl B, Cohen-Solal M, Aubry-Rozier B, Eriksen EF, Guanabens N, Obermayer-Pietsch B, Ralston SH, Eastell R, Zillikens MC. Discontinuation of Denosumab therapy for osteoporosis: A systematic review and position statement by ECTS. Bone. 2017 Dec;105:11-17. doi: 10.1016/j.bone.2017.08.003. Epub 2017 Aug 5. PMID 28789921
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Greene JG. A factor analytic study of climacteric symptoms. J Psychosom Res. 1976;20(5):425-30. doi: 10.1016/0022-3999(76)90005-2. No abstract available. PMID 1003364
- [Background] Derogatis LR, Rosen R, Leiblum S, Burnett A, Heiman J. The Female Sexual Distress Scale (FSDS): initial validation of a standardized scale for assessment of sexually related personal distress in women. J Sex Marital Ther. 2002 Jul-Sep;28(4):317-30. doi: 10.1080/00926230290001448. PMID 12082670
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Radtke JV, Terhorst L, Cohen SM. The Menopause-Specific Quality of Life Questionnaire: psychometric evaluation among breast cancer survivors. Menopause. 2011 Mar;18(3):289-95. doi: 10.1097/gme.0b013e3181ef975a. PMID 20881889
- [Background] Shieh A, Karlamangla AS, Gossiel F, Eastell R, Burnett-Bowie SA, Greendale GA. Estimating Net Bone Formation Relative to Resorption Using Reference Bone Turnover Markers. J Clin Endocrinol Metab. 2025 Jul 15;110(8):e2544-e2552. doi: 10.1210/clinem/dgae842. PMID 39657000
- [Background] Nathorst-Boos J, Floter A, Jarkander-Rolff M, Carlstrom K, Schoultz Bv. Treatment with percutanous testosterone gel in postmenopausal women with decreased libido--effects on sexuality and psychological general well-being. Maturitas. 2006 Jan 10;53(1):11-8. doi: 10.1016/j.maturitas.2005.01.002. Epub 2005 Sep 23. PMID 16183220
- [Background] Donovitz G, Cotten M. Breast Cancer Incidence Reduction in Women Treated with Subcutaneous Testosterone: Testosterone Therapy and Breast Cancer Incidence Study. Eur J Breast Health. 2021 Mar 31;17(2):150-156. doi: 10.4274/ejbh.galenos.2021.6213. eCollection 2021 Apr. PMID 33870115
- [Background] Glaser RL, York AE, Dimitrakakis C. Incidence of invasive breast cancer in women treated with testosterone implants: a prospective 10-year cohort study. BMC Cancer. 2019 Dec 30;19(1):1271. doi: 10.1186/s12885-019-6457-8. PMID 31888528
- [Background] Goldstat R, Briganti E, Tran J, Wolfe R, Davis SR. Transdermal testosterone therapy improves well-being, mood, and sexual function in premenopausal women. Menopause. 2003 Sep-Oct;10(5):390-8. doi: 10.1097/01.GME.0000060256.03945.20. PMID 14501599
- [Background] El-Hage G, Eden JA, Manga RZ. A double-blind, randomized, placebo-controlled trial of the effect of testosterone cream on the sexual motivation of menopausal hysterectomized women with hypoactive sexual desire disorder. Climacteric. 2007 Aug;10(4):335-43. doi: 10.1080/13697130701364644. PMID 17653960
- [Background] Simon J, Braunstein G, Nachtigall L, Utian W, Katz M, Miller S, Waldbaum A, Bouchard C, Derzko C, Buch A, Rodenberg C, Lucas J, Davis S. Testosterone patch increases sexual activity and desire in surgically menopausal women with hypoactive sexual desire disorder. J Clin Endocrinol Metab. 2005 Sep;90(9):5226-33. doi: 10.1210/jc.2004-1747. Epub 2005 Jul 12. PMID 16014407
- [Background] Panay N, Al-Azzawi F, Bouchard C, Davis SR, Eden J, Lodhi I, Rees M, Rodenberg CA, Rymer J, Schwenkhagen A, Sturdee DW. Testosterone treatment of HSDD in naturally menopausal women: the ADORE study. Climacteric. 2010 Apr;13(2):121-31. doi: 10.3109/13697131003675922. PMID 20166859
- [Background] Shifren JL, Davis SR, Moreau M, Waldbaum A, Bouchard C, DeRogatis L, Derzko C, Bearnson P, Kakos N, O'Neill S, Levine S, Wekselman K, Buch A, Rodenberg C, Kroll R. Testosterone patch for the treatment of hypoactive sexual desire disorder in naturally menopausal women: results from the INTIMATE NM1 Study. Menopause. 2006 Sep-Oct;13(5):770-9. doi: 10.1097/01.gme.0000243567.32828.99. PMID 16932240
- [Background] Hofling M, Lundstrom E, Azavedo E, Svane G, Hirschberg AL, von Schoultz B. Testosterone addition during menopausal hormone therapy: effects on mammographic breast density. Climacteric. 2007 Apr;10(2):155-63. doi: 10.1080/13697130701258812. PMID 17453864
- [Background] Fooladi E, Bell RJ, Jane F, Robinson PJ, Kulkarni J, Davis SR. Testosterone improves antidepressant-emergent loss of libido in women: findings from a randomized, double-blind, placebo-controlled trial. J Sex Med. 2014 Mar;11(3):831-9. doi: 10.1111/jsm.12426. Epub 2014 Jan 16. PMID 24433574
- [Background] Davis SR, Hirschberg AL, Wagner LK, Lodhi I, von Schoultz B. The effect of transdermal testosterone on mammographic density in postmenopausal women not receiving systemic estrogen therapy. J Clin Endocrinol Metab. 2009 Dec;94(12):4907-13. doi: 10.1210/jc.2009-1523. Epub 2009 Oct 22. PMID 19850682
- [Background] Davis SR, van der Mooren MJ, van Lunsen RH, Lopes P, Ribot C, Rees M, Moufarege A, Rodenberg C, Buch A, Purdie DW. Efficacy and safety of a testosterone patch for the treatment of hypoactive sexual desire disorder in surgically menopausal women: a randomized, placebo-controlled trial. Menopause. 2006 May-Jun;13(3):387-96. doi: 10.1097/01.gme.0000179049.08371.c7. PMID 16735935
- [Background] Buster JE, Kingsberg SA, Aguirre O, Brown C, Breaux JG, Buch A, Rodenberg CA, Wekselman K, Casson P. Testosterone patch for low sexual desire in surgically menopausal women: a randomized trial. Obstet Gynecol. 2005 May;105(5 Pt 1):944-52. doi: 10.1097/01.AOG.0000158103.27672.0d. PMID 15863529
- [Background] Kocoska-Maras L, Hirschberg AL, Bystrom B, Schoultz BV, Radestad AF. Testosterone addition to estrogen therapy - effects on inflammatory markers for cardiovascular disease. Gynecol Endocrinol. 2009 Dec;25(12):823-7. doi: 10.3109/09513590903056134. PMID 19906002
- [Background] Floter A, Nathorst-Boos J, Carlstrom K, Ohlsson C, Ringertz H, Schoultz Bv. Effects of combined estrogen/testosterone therapy on bone and body composition in oophorectomized women. Gynecol Endocrinol. 2005 Mar;20(3):155-60. doi: 10.1080/09513590400021193. PMID 16019355
- [Background] Floter A, Nathorst-Boos J, Carlstrom K, von Schoultz B. Addition of testosterone to estrogen replacement therapy in oophorectomized women: effects on sexuality and well-being. Climacteric. 2002 Dec;5(4):357-65. PMID 12626215
- [Background] Moller MC, Bartfai AB, Radestad AF. Effects of testosterone and estrogen replacement on memory function. Menopause. 2010 Sep-Oct;17(5):983-9. doi: 10.1097/gme.0b013e3181dc2e40. PMID 20555288
- [Background] Moller MC, Radestad AF, von Schoultz B, Bartfai A. Effect of estrogen and testosterone replacement therapy on cognitive fatigue. Gynecol Endocrinol. 2013 Feb;29(2):173-6. doi: 10.3109/09513590.2012.730568. Epub 2012 Oct 25. PMID 23095007
- [Background] Dias RS, Kerr-Correa F, Moreno RA, Trinca LA, Pontes A, Halbe HW, Gianfaldoni A, Dalben IS. Efficacy of hormone therapy with and without methyltestosterone augmentation of venlafaxine in the treatment of postmenopausal depression: a double-blind controlled pilot study. Menopause. 2006 Mar-Apr;13(2):202-11. doi: 10.1097/01.gme.0000198491.34371.9c. PMID 16645534
- [Background] Shifren JL, Braunstein GD, Simon JA, Casson PR, Buster JE, Redmond GP, Burki RE, Ginsburg ES, Rosen RC, Leiblum SR, Caramelli KE, Mazer NA. Transdermal testosterone treatment in women with impaired sexual function after oophorectomy. N Engl J Med. 2000 Sep 7;343(10):682-8. doi: 10.1056/NEJM200009073431002. PMID 10974131
- [Background] Wisniewski AB, Nguyen TT, Dobs AS. Evaluation of high-dose estrogen and high-dose estrogen plus methyltestosterone treatment on cognitive task performance in postmenopausal women. Horm Res. 2002;58(3):150-5. doi: 10.1159/000064491. PMID 12218381
- [Background] Penteado SR, Fonseca AM, Bagnoli VR, Abdo CH, Junior JM, Baracat EC. Effects of the addition of methyltestosterone to combined hormone therapy with estrogens and progestogens on sexual energy and on orgasm in postmenopausal women. Climacteric. 2008 Feb;11(1):17-25. doi: 10.1080/13697130701741932. PMID 18202961
- [Background] Leao LM, Duarte MP, Silva DM, Bahia PR, Coeli CM, de Farias ML. Influence of methyltestosterone postmenopausal therapy on plasma lipids, inflammatory factors, glucose metabolism and visceral fat: a randomized study. Eur J Endocrinol. 2006 Jan;154(1):131-9. doi: 10.1530/eje.1.02065. PMID 16382002
- [Background] de Paula FJ, Soares JM Jr, Haidar MA, de Lima GR, Baracat EC. The benefits of androgens combined with hormone replacement therapy regarding to patients with postmenopausal sexual symptoms. Maturitas. 2007 Jan 20;56(1):69-77. doi: 10.1016/j.maturitas.2006.06.005. Epub 2006 Jul 5. PMID 16822626
- [Background] Basaria S, Nguyen T, Rosenson RS, Dobs AS. Effect of methyl testosterone administration on plasma viscosity in postmenopausal women. Clin Endocrinol (Oxf). 2002 Aug;57(2):209-14. doi: 10.1046/j.1365-2265.2002.01584.x. PMID 12153599
- [Background] Islam RM, Bell RJ, Green S, Page MJ, Davis SR. Safety and efficacy of testosterone for women: a systematic review and meta-analysis of randomised controlled trial data. Lancet Diabetes Endocrinol. 2019 Oct;7(10):754-766. doi: 10.1016/S2213-8587(19)30189-5. Epub 2019 Jul 25. PMID 31353194
- [Background] Bowen RL, Perry G, Xiong C, Smith MA, Atwood CS. A clinical study of lupron depot in the treatment of women with Alzheimer's disease: preservation of cognitive function in patients taking an acetylcholinesterase inhibitor and treated with high dose lupron over 48 weeks. J Alzheimers Dis. 2015;44(2):549-60. doi: 10.3233/JAD-141626. PMID 25310993
- [Background] Ludvigsson JF, Adolfsson J, Hoistad M, Rydelius PA, Kristrom B, Landen M. A systematic review of hormone treatment for children with gender dysphoria and recommendations for research. Acta Paediatr. 2023 Nov;112(11):2279-2292. doi: 10.1111/apa.16791. Epub 2023 May 1. PMID 37069492
- [Background] Glaser R, York AE, Dimitrakakis C. Beneficial effects of testosterone therapy in women measured by the validated Menopause Rating Scale (MRS). Maturitas. 2011 Apr;68(4):355-61. doi: 10.1016/j.maturitas.2010.12.001. Epub 2010 Dec 21. PMID 21177051
- [Background] Chidi-Ogbolu N, Baar K. Effect of Estrogen on Musculoskeletal Performance and Injury Risk. Front Physiol. 2019 Jan 15;9:1834. doi: 10.3389/fphys.2018.01834. eCollection 2018. PMID 30697162
- [Background] Greendale GA, Sternfeld B, Huang M, Han W, Karvonen-Gutierrez C, Ruppert K, Cauley JA, Finkelstein JS, Jiang SF, Karlamangla AS. Changes in body composition and weight during the menopause transition. JCI Insight. 2019 Mar 7;4(5):e124865. doi: 10.1172/jci.insight.124865. eCollection 2019 Mar 7. PMID 30843880
- [Background] Juel Mortensen L, Kooij I, Lorenzen M, Rye Jorgensen N, Roder A, Jorgensen A, Andersson AM, Juul A, Blomberg Jensen M. Injection of luteinizing hormone or human chorionic gonadotropin increases calcium excretion and serum PTH in males. Cell Calcium. 2024 Sep;122:102908. doi: 10.1016/j.ceca.2024.102908. Epub 2024 May 24. PMID 38852333
- [Background] Neff LM, Hoffmann ME, Zeiss DM, Lowry K, Edwards M, Rodriguez SM, Wachsberg KN, Kushner R, Landsberg L. Core body temperature is lower in postmenopausal women than premenopausal women: potential implications for energy metabolism and midlife weight gain. Cardiovasc Endocrinol. 2016 Dec;5(4):151-154. doi: 10.1097/XCE.0000000000000078. PMID 28111609
- [Background] van Gastel P, van der Zanden M, Telting D, Filius M, Bancsi L, de Boer H. Luteinizing hormone-releasing hormone receptor antagonist may reduce postmenopausal flushing. Menopause. 2012 Feb;19(2):178-85. doi: 10.1097/gme.0b013e31822542ca. PMID 21926922
- [Background] Casper RF, Yen SS. Neuroendocrinology of menopausal flushes: an hypothesis of flush mechanism. Clin Endocrinol (Oxf). 1985 Mar;22(3):293-312. doi: 10.1111/j.1365-2265.1985.tb03243.x. No abstract available. PMID 3884189
- [Background] Manson JE, Chlebowski RT, Stefanick ML, Aragaki AK, Rossouw JE, Prentice RL, Anderson G, Howard BV, Thomson CA, LaCroix AZ, Wactawski-Wende J, Jackson RD, Limacher M, Margolis KL, Wassertheil-Smoller S, Beresford SA, Cauley JA, Eaton CB, Gass M, Hsia J, Johnson KC, Kooperberg C, Kuller LH, Lewis CE, Liu S, Martin LW, Ockene JK, O'Sullivan MJ, Powell LH, Simon MS, Van Horn L, Vitolins MZ, Wallace RB. Menopausal hormone therapy and health outcomes during the intervention and extended poststopping phases of the Women's Health Initiative randomized trials. JAMA. 2013 Oct 2;310(13):1353-68. doi: 10.1001/jama.2013.278040. PMID 24084921
- [Background] Collaborative Group on Hormonal Factors in Breast Cancer. Type and timing of menopausal hormone therapy and breast cancer risk: individual participant meta-analysis of the worldwide epidemiological evidence. Lancet. 2019 Sep 28;394(10204):1159-1168. doi: 10.1016/S0140-6736(19)31709-X. Epub 2019 Aug 29. PMID 31474332
- [Background] Monteleone P, Mascagni G, Giannini A, Genazzani AR, Simoncini T. Symptoms of menopause - global prevalence, physiology and implications. Nat Rev Endocrinol. 2018 Apr;14(4):199-215. doi: 10.1038/nrendo.2017.180. Epub 2018 Feb 2. PMID 29393299
- [Background] Vestergaard P, Rejnmark L, Mosekilde L. Increased mortality in patients with a hip fracture-effect of pre-morbid conditions and post-fracture complications. Osteoporos Int. 2007 Dec;18(12):1583-93. doi: 10.1007/s00198-007-0403-3. Epub 2007 Jun 14. PMID 17566814
- [Background] Compston JE, McClung MR, Leslie WD. Osteoporosis. Lancet. 2019 Jan 26;393(10169):364-376. doi: 10.1016/S0140-6736(18)32112-3. PMID 30696576
- [Background] Grey A, Bolland MJ. The effect of treatments for osteoporosis on mortality. Osteoporos Int. 2013 Jan;24(1):1-6. doi: 10.1007/s00198-012-2176-6. Epub 2012 Oct 18. PMID 23076683
- [Background] Lee E, Anselmo M, Tahsin CT, Vanden Noven M, Stokes W, Carter JR, Keller-Ross ML. Vasomotor symptoms of menopause, autonomic dysfunction, and cardiovascular disease. Am J Physiol Heart Circ Physiol. 2022 Dec 1;323(6):H1270-H1280. doi: 10.1152/ajpheart.00477.2022. Epub 2022 Nov 11. PMID 36367692
- [Background] Wright NC, Looker AC, Saag KG, Curtis JR, Delzell ES, Randall S, Dawson-Hughes B. The recent prevalence of osteoporosis and low bone mass in the United States based on bone mineral density at the femoral neck or lumbar spine. J Bone Miner Res. 2014 Nov;29(11):2520-6. doi: 10.1002/jbmr.2269. PMID 24771492
- [Background] Knight MG, Anekwe C, Washington K, Akam EY, Wang E, Stanford FC. Weight regulation in menopause. Menopause. 2021 May 24;28(8):960-965. doi: 10.1097/GME.0000000000001792. PMID 34033603
- [Background] Woods NF, Mitchell ES. Symptoms during the perimenopause: prevalence, severity, trajectory, and significance in women's lives. Am J Med. 2005 Dec 19;118 Suppl 12B:14-24. doi: 10.1016/j.amjmed.2005.09.031. PMID 16414323
- [Background] Nelson HD. Menopause. Lancet. 2008 Mar 1;371(9614):760-70. doi: 10.1016/S0140-6736(08)60346-3. PMID 18313505